CLINICAL TRIAL: NCT03464110
Title: Communication Coaching to Improve Patient and Clinician Satisfaction in Cardiology Encounters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00091691
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Improved Communication Between Clinician and Patient

STUDY DESIGN:
Intervention Model Description: Interventional: To determine the effect of a clinician communication coaching intervention versus control on an objective measure of the quality of communication (primary outcome) and patients' perceptions of the quality of patient-centered care (secondary outcome), both overall and within Black and White patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Investigator will compare patients randomized into the intervention group to those who receive standard of care.
- Communication Intervention (Experimental): The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
  Interventions: Behavioral: Communication Intervention

INTERVENTIONS:
Behavioral: Communication Intervention — . The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
  Arms: Communication Intervention

SUMMARY:
The purpose of this study is to determine the effect of a clinician communication coaching intervention versus control on an objective measure of the quality of communication (primary outcome) and patients' perceptions of the quality of patient-centered care (secondary outcome), both overall and within Black and White patients.

DETAILED DESCRIPTION:
The investigators propose a two-arm cluster randomized controlled design, in which the unit of randomization is the clinician. Up to fifty cardiology clinicians will be randomly assigned to either the coaching intervention or to a control condition. The investigators will recruit up to 50 clinicians to ensure that we have at least 40 clinicians with complete pre- and post-intervention measures. Although the unit of randomization is the clinician, the unit of evaluation is the patient: 10 patients per clinician who get cardiology care from the enrolled clinicians will consent to audio-recording of their encounters and to completing the surveys. Clinicians randomized to the intervention will obtain verbal consent from additional patients to audio-record the encounter for coaching. The intervention will be delivered in the clinic or via video-conference (Skype or Facetime), providing individual coaching and professional feedback on the communication behaviors encounters. The investigators will also measure Press Ganey scores by clinician pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older
* Must be able to read
* Must speak English
* Capable of providing informed consent
* Must be receiving continuity care from and enrolled clinician

Exclusion Criteria:

* Currently hospitalized
* Awaiting heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Pollak, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Duke University Medical Center - Cancer Prevention, Detection and Control, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollak KI, Olsen MK, Yang H, Prose N, Jackson LR 2nd, Pinheiro SO, Dunbar TK, Johnson KS. Effect of a Coaching Intervention to Improve Cardiologist Communication: A Randomized Clinical Trial. JAMA Intern Med. 2023 Jun 1;183(6):544-553. doi: 10.1001/jamainternmed.2023.0629. PMID 37036721

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care - Physicians; Standard of Care - Patients: Investigator will compare patients randomized into the intervention group to those who receive standard of care.
- Communication Intervention - Physicians; Communication Intervention - Patients: The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
  Communication Intervention: . The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
Period: Overall Study
Arm/Group | Standard of Care - Physicians | Communication Intervention - Physicians | Standard of Care - Patients | Communication Intervention - Patients
Started | 20 | 20 | 120 | 120
Completed | 20 | 20 | 120 | 120
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care (Provider): Control cardiology providers. Receiving no intervention.
- Communication Intervention (Provider): The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
  Communication Intervention: . The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
- Standard of Care (Patient): Patients seen by standard of care (control) cardiology providers.
- Communication Intervention (Patient): Patients seen by cardiologists who received the communication coaching intervention.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Provider) | Communication Intervention (Provider) | Standard of Care (Patient) | Communication Intervention (Patient) | Total
Number analyzed (Participants) | 20 | 20 | 120 | 120 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9) | 46 (9) | 60 (14) | 56 (15) | 56.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 65 | 61 | 133
  Male | 16 | 17 | 55 | 59 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 5
  Not Hispanic or Latino | 18 | 19 | 119 | 119 | 275
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 4 | 0 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 60 | 58 | 120
  White | 9 | 16 | 60 | 62 | 147
  More than one race | 3 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Average Number of Direct Patient Care Hours per Week [Mean (Standard Deviation); unit: hours per week] — Population: Only applicable to Providers. This data was not collected for patients - not applicable.
  hours per week
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 40
    (all) | 32 (14) | 29 (15) |  |  | 30 (15)
Type of visit [Count of Participants; unit: Participants] — Procedural versus non-procedural Population: Only applicable to Providers. This data was not collected for patients - not applicable.
  Participants
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 40
    Procedural | 7 | 8 |  |  | 15
    Non-procedural | 13 | 12 |  |  | 25
No prior communication training [Count of Participants; unit: Participants] — Population: Only applicable to Providers. This data was not collected for patients - not applicable.
  Participants
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 40
    (all) | 13 | 14 |  |  | 27
Practice Specialty [Count of Participants; unit: Participants] — Population: Only applicable to Providers. This data was not collected for patients - not applicable.
  Participants
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 40
    General | 8 | 6 |  |  | 14
    Electrophysiology | 3 | 4 |  |  | 7
    Interventional | 4 | 3 |  |  | 7
    Advanced Heart Failure | 3 | 5 |  |  | 8
    Cardiac Imaging | 2 | 1 |  |  | 3
    Congenital disease | 0 | 1 |  |  | 1
Years in Practice [Count of Participants; unit: Participants] — Population: Only applicable to Providers. This data was not collected for patients - not applicable.
  Participants
    number analyzed (Participants) | 20 | 20 | 0 | 0 | 40
    Less than a Year | 1 | 0 |  |  | 1
    1-5 Years | 3 | 0 |  |  | 3
    6-10 Years | 2 | 5 |  |  | 7
    11-15 Years | 3 | 6 |  |  | 9
    More than 15 Years | 11 | 9 |  |  | 20
    Prefer not to answer | 0 | 0 |  |  | 0
Patient Education [Count of Participants; unit: Participants] — Population: Only applicable to Patients. This data was not collected for providers - not applicable.
  Participants
    Eighth Grade or Less: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Eighth Grade or Less |  |  | 1 | 0 | 1
    Some High School. Completed high school or GED.: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Some High School. Completed high school or GED. |  |  | 24 | 29 | 53
    Vocational or trade school: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Vocational or trade school |  |  | 8 | 7 | 15
    Some college or university but no degree: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Some college or university but no degree |  |  | 24 | 15 | 39
    Associate's degree from college or university: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Associate's degree from college or university |  |  | 13 | 10 | 23
    Bachelor's degree: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Bachelor's degree |  |  | 21 | 25 | 46
    Some graduate or professional school: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Some graduate or professional school |  |  | 6 | 2 | 8
    Graduate or professional degree: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Graduate or professional degree |  |  | 20 | 28 | 48
    Missing: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Missing |  |  | 3 | 4 | 7
Patient Marital Status [Count of Participants; unit: Participants] — Married or live with partner. Population: Only applicable to Patients. This data was not collected for providers - not applicable.
  Participants
    number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    (all) |  |  | 73 | 66 | 139
Patient Employment [Count of Participants; unit: Participants] — Working full or part time. Population: Only applicable to Patients. This data was not collected for providers - not applicable.
  Participants
    number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    (all) |  |  | 42 | 43 | 85
Patient Insurance [Count of Participants; unit: Participants] — Population: Only applicable to Patients. This data was not collected for providers - not applicable.
  Participants
    Plan purchased via employer or union: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Plan purchased via employer or union |  |  | 40 | 49 | 89
    Plan, self or family purchased: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Plan, self or family purchased |  |  | 2 | 4 | 6
    Medicare: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Medicare |  |  | 57 | 38 | 95
    Medicaid: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Medicaid |  |  | 11 | 16 | 27
    TRICARE: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    TRICARE |  |  | 2 | 6 | 8
    Some other source: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Some other source |  |  | 3 | 1 | 4
    None: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    None |  |  | 2 | 2 | 4
    Missing: number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    Missing |  |  | 3 | 4 | 7
Patient Income [Count of Participants; unit: Participants] — Population: Only applicable to Patients. This data was not collected for providers - not applicable.
  Participants
    number analyzed (Participants) | 0 | 0 | 120 | 120 | 240
    After paying the bills, you still have enough money for special things that you want |  |  | 61 | 56 | 117
    You have enough money to pay the bills, but little spare money to buy extra or special things |  |  | 36 | 33 | 69
    You have money to pay the bills, but only because you have cut back on things |  |  | 10 | 8 | 18
    You are having difficulty paying the bills, no matter what you do |  |  | 6 | 6 | 12
    Prefer not to answer |  |  | 4 | 13 | 17
    Missing |  |  | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cardiologist Behavior as Measured by WISER (Writing, Immersive Experiences, Speaking, Ethical Communication, and Research) Assessment.
Description: WISER is based on established codebooks (i.e., Motivational Interviewing Treatment Integrity manual, and Suchman's codebook for patient emotion and physician empathic responses). Communication coaches taught five skills: 1) sitting down and making eye contact with all in the room, 2) open-ended questions, 3) reflective statements, 4) empathic statements, and 5) "What questions do you have?". Reported here is the number of Reflective Statements made.
Time Frame: One encounter, up to approximately 1 hour
Population: Only applies to Patient groups. Data not collected on 10 participants.
Measure: Mean (Standard Deviation); unit: Number of Reflective Statements
Groups:
- Communication Intervention - Patients: The intervention will contain elements of Motivational Interviewing coaching but also will teach providers how to address patient emotion and increase the efficiency of their visits. Clinicians randomized to the intervention will receive a tailored communication coaching intervention that includes didactic elements, audio recording encounters and providing feedback, and role-playing.
Arm/Group | Standard of Care - Patients | Communication Intervention - Patients
Number analyzed (Participants) | 113 | 117
Number of Reflective Statements | 11.95 (8.81) | 13.15 (9.96)

2. Primary Outcome: Cardiologist Behavior as Measured by WISER (Writing, Immersive Experiences, Speaking, Ethical Communication, and Research) Assessment.
Description: WISER is based on established codebooks (i.e., Motivational Interviewing Treatment Integrity manual, and Suchman's codebook for patient emotion and physician empathic responses). Communication coaches taught five skills: 1) sitting down and making eye contact with all in the room, 2) open-ended questions, 3) reflective statements, 4) empathic statements, and 5) "What questions do you have?". Reported here is the number of Open-ended Questions asked.
Time Frame: One encounter, up to approximately 1 hour
Population: Only applies to Patient groups. Data not collected on 10 participants.
Measure: Mean (Standard Deviation); unit: questions asked
Arm/Group | Standard of Care - Patients | Communication Intervention - Patients
Number analyzed (Participants) | 113 | 117
questions asked | 3.41 (2.84) | 3.28 (2.89)

3. Primary Outcome: Ratio of Empathic Responses to Empathic Opportunities
Description: Communication coaches taught five skills: 1) sitting down and making eye contact with all in the room, 2) open-ended questions, 3) reflective statements, 4) empathic statements, and 5) "What questions do you have?". Reported here is the ratio of empathic responses to empathic opportunities.
Time Frame: One encounter, up to approximately 1 hour
Population: Participants with encounters in which the clinician had at least one empathic response. Only applies to Patient groups.
Measure: Mean (Standard Deviation); unit: ratio of responses to opportunities
Arm/Group | Standard of Care - Patients | Communication Intervention - Patients
Number analyzed (Participants) | 35 | 48
ratio of responses to opportunities | 0.20 (0.36) | 0.50 (0.47)

4. Secondary Outcome: Global Ratings of Communication as Measured by WISER (Writing, Immersive Experiences, Speaking, Ethical Communication, and Research) Assessment
Description: Global ratings represent areas of effective communication that address many domains of patient-centered communication or areas that facilitate patient satisfaction with communication. WISER is based on established codebooks (i.e., Motivational Interviewing Treatment Integrity manual, and Suchman's codebook for patient emotion and physician empathic responses. Scores of 1-5 with 3 being average, 1 being below average, 5 being above average.
Time Frame: One encounter, up to approximately 1 hour
Population: Only applies to Patient groups. Data not collected on 10 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care - Patients | Communication Intervention - Patients
Number analyzed (Participants) | 113 | 117
score on a scale
  Attentiveness | 3.8 (0.9) | 3.8 (0.9)
  Flow | 2.9 (1.1) | 3.3 (1.0)
  Concern | 4.0 (0.8) | 4.2 (0.7)
  Respect | 3.8 (1.0) | 4.0 (0.9)
  Warmth | 3.5 (0.9) | 3.6 (0.8)

ADVERSE EVENTS:
Time Frame: One encounter, up to approximately 1 hour
Groups:
- Standard of Care (Provider): Investigator will compare patients randomized into the intervention group to those who receive standard of care.
- Standard of Care (Patient): Patients seen by Standard of Care cardiologists
- Communication Intervention (Patient): Patients seen by Communication Intervention cardiologists
Arm/Group | Standard of Care (Provider) | Communication Intervention (Provider) | Standard of Care (Patient) | Communication Intervention (Patient)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03464110/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03464110/SAP_001.pdf
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03464110/ICF_002.pdf